CLINICAL TRIAL: NCT06435598
Title: Effect of Video-Based Health Education Intervention on Insulin Therapy Among Adults With Diabetes Mellitus in Dhulikhel Hospital: A Randomized Controlled Trial This Research Aims to Investigate the Effectiveness of Video-based Health Education in Supporting Insulin Therapy in Diabetes Mellitus Patients Visiting Dhulikhel Hospital. With the Increasing Patients With Insulin Therapy and the Need for Effective Patient Education, it is Essential to Evaluate the Impact of Video-based Educational Interventions Specifically Tailored for Patients Undergoing Insulin Therapy.
Brief Title: Tittle: Effect of Video-Based Health Education Intervention on Insulin Therapy Among Adults With Diabetes Mellitus in Dhulikhel Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Subina Manandhar, Assistant Professor in Nursing Department, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 737/2023
Record Dates: First submitted 2024-05-15; First posted 2024-05-30 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Knowledge on Insulin Therapy; Practice on Insulin Administration
Keywords: Diabetes mellitus; Educational Video on insulin therapy; Insulin Therapy for diabetes mellitus; Knowledge on insulin therapy; Practice on insulin administration; Usual Care on insulin administration
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is an open-label two-arm randomized trial. Investigator will allocate half of the participants to the video-based health education and usual care, while the other half of the participants will receive usual care only. (Fig 1) Randomization: Block randomization will be done to allocate adults to intervention or usual care group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Educational video and usual care) (Experimental): Investigator will allocate sixty- three of the participants to the video-based health education and usual care
  Interventions: Other: video-based health education
- Control Group (Usual Care) (No Intervention): Investigator will allocate sixty-three of the participants to usual care only

INTERVENTIONS:
Other: video-based health education — The video- based health education program guided by the Health Belief Model will be designed to provide tailored information on insulin therapy in diabetes. Health Belief Model(HBM) emphasizes changes in people's behavior are acquired through awareness of risk factors and perceived health benefits. The video will provide general information on insulin, types of insulin, its administration technique and storage.
  Other Names: Usual Care
  Arms: Intervention Group (Educational video and usual care)

SUMMARY:
Insulin is an essential therapy for treating diabetes, but many patients lack standard insulin injection skills. Learning the method of proper insulin injection technique is crucial for diabetes patients as it promotes treatment compliance, ensures safety, improves treatment efficacy, and contributes to better overall health outcomes. Adequate training and understanding of the proper technique enhance patient self-efficacy and empower them to take an active role in managing their diabetes mellitus. It empowers patients to effectively manage their diabetes and maintain optimal blood glucose control, ultimately leading to a better quality of life. This research aims to investigate the effectiveness of video-based health education in supporting insulin therapy in diabetes mellitus patients visiting Dhulikhel Hospital. With the increasing patients with insulin therapy and the need for effective patient education, it is essential to evaluate the impact of video-based educational interventions specifically tailored for patients undergoing insulin therapy. A randomized control trial method will be used for the study. Participants will be randomly assigned to either an experimental group receiving face to face educational session with video-based education or a control group receiving standard face-to-face educational session. Data will be collected through pre and post intervention assessments. The study's outcomes will help optimize patient care, increase accessibility to healthcare services and potentially reshape the way insulin therapy is delivered to Diabetes Mellitus patients.

DETAILED DESCRIPTION:
Background:

The prevalence of diabetes is high, and is expected to increase in developing countries or regions such as China, India, Brazil and Southeast Asia. Diabetes Mellitus is a chronic condition that requires lifelong management insulin therapy being a crucial component for many patients. Proper understanding and adherence to insulin are essential for achieving optimal health outcomes. Patient education plays a vital role in enhancing knowledge, self-management skills, and treatment adherence. Video- based health education offers several advantages including accessibility, flexibility and the ability to provide visual demonstrations. It can empower patients to actively participate in their self-care and improve their overall well-being.

Proper injection technique ensures the safe and effective delivery of insulin into the body. This helps minimize the risk of complications such as infections, bruising, discomfort, pain and incorrect dosage administration. Proper injection depth, angle and site rotation contribute to consistent absorption of insulin, leading better blood glucose control. This is possible when patients are confident in their ability to administer insulin correctly with the right training and education.

Overall, this study holds significant importance as it addresses the gap in knowledge regarding the effectiveness of video-based health education in supporting insulin therapy for Diabetes Mellitus patients. Its findings will have implication for optimizing patient education strategies, enhancing treatment adherence and ultimately improving the quality of life for individuals living with Diabetes Mellitus.

Rational/justification:

By conducting this randomized controlled trial, Investigator aim to contribute to the patient education in diabetes management. It will help to optimize patient education methods, enhance treatment adherence and ultimately lead to better health outcomes for Diabetes mellitus patients on insulin therapy.

General Objective:

To explore whether the use of video-based health education program results in better knowledge, practice of insulin therapy technique when compared to usual care among adults with diabetes mellitus in Dhulikhel Hospital.

Specific Objective:

* To determine video-based health education program compared with usual care improves the practice score of insulin therapy technique among adults with diabetes mellitus in Dhulikhel Hospital.
* To find out video-based health education program compared with usual care increases the knowledge score of insulin therapy technique among adults with diabetes mellitus in Dhulikhel Hospital.
* To find out the association of practice of insulin therapy technique before the intervention with selected socio demographic variable.

Research Hypothesis Video-based health education intervention improves knowledge and practice of insulin therapy technique among adults with diabetes mellitus attending Dhulikhel Hospital.

Study Variables:

Dependent Variables: Knowledge and Practice in Insulin Therapy Independent Variables: Socio Demography Data, Educational Video Intervention

Research Method:

Quantitative

This is an open-label two-arm randomized trial. Investigator will allocate half of the participants to the video-based health education and usual care, while the other half of the participants will receive usual care only. (Fig 1) Randomization: Block randomization will be done to allocate adults to intervention or usual care group. A random sequence number will be generated in blocks of size of ten using STATA 14 by a statistician. The random numbers will be copied in an excel form and median will be calculated for each block. The numbers below the median will be assigned as 'usual care group' and the numbers above the median will be assigned as 'intervention group'. Diabetic nurses and other nursing staff at the medical OPD and ward in Dhulikhel hospital will identify adults with diabetes and will check their eligibility. Investigator will explain ethical considerations, the importance of maintaining confidentiality during the research process, the voluntary nature of the participation, and the option to quit the study at any time. Investigator will enroll adults providing consent. After taking written consent, investigator will interview adults for baseline characteristics and their knowledge on insulin therapy. The interview will take 30-35 minutes.

Allocation concealment: A computer-based program will randomly allocate participants to either video-based education plus usual care or in a group with usual care only. Block randomization will be done to allocate adults to intervention or usual care group. A random sequence number will be generated in blocks of size of ten using STATA 14 by a statistician. The random numbers will be copied in an excel form and median will be calculated for each block. The numbers below the median will be assigned as 'usual care group' and the numbers above the median will be assigned as 'intervention group'. For randomization, the participants who have agreed to participate will be randomized into either the intervention or control group, with a 1:1 ratio based on allocation sequence. The allocation sequence will be concealed from the research nurse and participants using sequentially numbered opaque sealed envelopes (SNOSE) method. The principal investigator will provide the sealed envelopes to the research nurse who will then assign participants' to the intervention. The participants, the service provider, and the research nurse will be aware of the intervention.

Intervention: The video-based health education program guided by the Health Belief Model will be designed to provide tailored information on insulin therapy in diabetes. Health Belief Model(HBM) emphasizes changes in people's behavior are acquired through awareness of risk factors and perceived health benefits. The video will provide general information on insulin, types of insulin, its administration technique and storage.

Usual Care: Both intervention and control group will receive the usual standard diabetic care from Dhulikhel hospital which includes diabetic counseling, health teachings, etc.

ELIGIBILITY:
Inclusion Criteria:

* Adult more than or equal to 18 years.
* Adult diagnosed with diabetes mellitus
* Adult under insulin therapy
* Adult owns smartphone with social media account

Exclusion Criteria:

* Patient with learning difficulties (dementia), hearing or visual impairment and hand tremors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge on insulin therapy | 4 months
  Knowledge on insulin therapy will cover structured questionnaire
Practice of insulin administration technique | 4 months
  Practice of insulin administration will be assessed by checklist

CONTACTS AND LOCATIONS:
Overall Officials: Subina Manandhar, M.Sc., Principal Investigator — Kathmandu University School of Medical Sciences; Kunta D Pun, PhD, Study Director — Kathmandu University School of Medical Sciences
Locations (1):
- Dhulikhel Hospital, Dhulikhel, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cui M, Wu X, Mao J, Wang X, Nie M (2016) T2DM Self-Management via Smartphone Applications: A Systematic Review and Meta-Analysis. PLOS ONE 11(11): e0166718 — https://doi.org/10.1371/journal.pone.0166718
- See also: 12. Frid AH, Kreugel G, Grassi G, Halimi S, Hicks D, Hirsch LJ, et al. New Insulin Delivery Recommendations. Mayo Clin Proc [Internet]. 2016;91(9):1231-55 — http://dx.doi.org/10.1016/j.mayocp.2016.06.010